CLINICAL TRIAL: NCT04205435
Title: a Safety and Efficacy Study of β-globin Restored Autologous Hematopoietic Stem Cells for β-thalassemia Major Patients With CVS-654 Mutation
Brief Title: β-globin Restored Autologous HSC in β-thalassemia Major Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bioray Laboratories (Industry)
Collaborators: The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-BRL-00CH2
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-09

CONDITIONS: β-thalassemia Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- β-globin restored autologous HSC (Experimental): each subject will accept one dose of β-globin restored autologous hematopoietic stem cells
  Interventions: Biological: β-globin restored autologous HSC

INTERVENTIONS:
Biological: β-globin restored autologous HSC — gene edited autologous hematopoietic stem cells with β-globin restoration

SUMMARY:
This is a single center, single arm, open-label study to determine the safety and efficacy of β-globin restored autologous hematopoietic stem cells in β- thalassemia major patients with CVS-654 mutation.

DETAILED DESCRIPTION:
β-globin restored autologous hematopoietic stem cells will be manufactured using CRISPR/Cas9 gene editing system. Subject participation for this study will be 1 year. Subjects who enroll in this study will be asked to participate in a subsequent long-term follow up study that will monitor the safety and efficacy of the treatment they receive for up to 15 years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* 5-15 years old. Clinically diagnosed as β-thalassemia major with IVS-654 gene mutation phenotype;
* Subjects or at least one legal guardian/agent understand and voluntarily sign informed consent.
* Subjects with no affection with EBV, HIV, CMV, TP, HAV, HBV and HCV.
* Subjects body condition eligible for autologous stem cell transplant.

Exclusion Criteria:

- Subjects acceptable for allogeneic hematopoietic stem cell transplantation and have an available fully matched related donor.

Active bacterial, viral, or fungal infection. Treated with erythropoietin prior 3 months. Immediate family member with any known hematological tumor. Subjects with severe psychiatric disorders to be unable to cooperate. Recently diagnosed as malaria. History of complex autoimmune disease. Persistent aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin value >3 x the upper limit of normal (ULN).

Subjects with severe heart, lung and kidney diseases. With serious iron overload. Any other condition that would render the subject ineligible for HSCT, as determined by the attending transplant physician or Investigator.

Subjects who are receiving treatment from another clinical study, or have received another gene therapy.

Subjects or guardians had resisted the guidance of the attending doctor. Subjects whom the investigators do not consider appropriate for participating in this clinical study.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with engraftment; | up to 42 days post transplant
Incidence and severity of adverse events as a measure of safety and tolerability. Adverse events assessed according to NCI-CTCAE v5.0 criteria | up to 60 days post transplant

SECONDARY OUTCOMES:
Proportion of subjects achieving transfusion independence; | up to 24 months post transplant
Proportion of subjects with a > = 50% reduced annualized volume of packed RBC transfusions. | up to 24 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Zhang, Prof, Principal Investigator — The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army
Locations (1):
- Shanghai Bioraylaboratory Inc, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brusson M, Miccio A. Genome editing approaches to beta-hemoglobinopathies. Prog Mol Biol Transl Sci. 2021;182:153-183. doi: 10.1016/bs.pmbts.2021.01.025. Epub 2021 Mar 1. PMID 34175041